CLINICAL TRIAL: NCT02622906
Title: Randomized Phase II Trial Evaluating the Efficiency of Pasireotide for the Treatment of Gastrointestinal Angiodysplasia in Endoscopic Treatment Failure
Brief Title: Pasireotide for the Treatment of Gastrointestinal Angiodysplasia in Endoscopic Treatment Failure
Acronym: ANGIOPAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Benamouzig (Other)
Responsible Party: Sponsor-Investigator, Robert Benamouzig, Professor, Hospital Avicenne
Organization: Hospital Avicenne (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-002579-40
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Angiodysplasia
Keywords: Gastrointestinal angiodysplasia; Pasireotide; Gastrointestinal bleeding
MeSH Terms: conditions — Angiodysplasia; Gastrointestinal Hemorrhage | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 1 injection per month during 6 months of the placebo product
  Interventions: Drug: Placebo
- Pasireotide (Active Comparator): 1 injection per month during 6 months of the Pasireotide LP (60mg/injection)
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide — 60 mg per month of the Pasireotide during 6 months
  Arms: Pasireotide
Drug: Placebo — Vehicule injection per month during 6 months
  Arms: Placebo

SUMMARY:
The angiodysplasias may be responsible for recurrent gastrointestinal bleeding and in some cases bleeding remaining inaccessible to endoscopic treatment. Several observational studies suggest that treatment with somatostatin analogue would reduce transfusion requirements in patients with recurrent bleeding due to angiodysplasia.

No randomized studies are available. The main objective of this study multicenter, prospective, randomized, was to assess the transfusion requirements in patients with recurrent bleeding due to angiodysplasia treated by a new analogue of somatostatin, Pasireotide, versus placebo.

Patients with recurrent gastrointestinal bleeding related to angiodysplasias, endoscopic treatment failure, with a need transfusion at least 6 red blood cells during the 6 months prior to inclusion could be randomized to receive monthly intramuscular injection of Pasireotide 60 mg or placebo for a period of 6 months. Patients were then followed for an additional 6 months after stopping treatment. A test monthly clinical and laboratory was performed during the six months of treatment then quarterly during the six months of surveillance.

DETAILED DESCRIPTION:
The angiodysplasias are abnormal communications between dilated capillaries and veins. Their presence in the digestive tract is probably due to venous obstruction associated with smooth muscle contractions. These vascular malformations are not a particularly significant cause of bleeding in elderly patients. The angiodysplasias are responsible for about 1% of upper gastrointestinal bleeding and up to 6% of the lower bleeding. However in case of gastrointestinal bleeding obscures the presence of angiodysplasia was found in 23% of cases through an exploration of the small intestine endoscopic video capsule enteroscopy or double balloon. Some conditions promote the development of angiodysplasias such as kidney failure with a prevalence of 13% in case of bleeding or cirrhosis. The responsibility of aortic stenosis is debated and could be a chance association. On the other hand, are more symptomatic bleeding in case of bleeding disorders, in particular von Willebrand disease.

The first line treatment is based on the destruction of endoscopic lesions by laser, or argon plasma coagulation electrocoagulation. However, these lesions may be inaccessible to endoscopic treatment, when they are too numerous or if patients with severe comorbidities, indicating against invasive endoscopic treatments. Iterative transfusions remain the only possible treatment for a significant proportion of patient which induces frequent hospitalizations, complications related to transfusions and a significant cost.

Hormonal treatments have been tried without success to prevent rebleeding. Anti-angiogenic as thalidomide have been tested in phase II trials in low number of the patients.

Somatostatin is a cyclic peptide secreted by D cells in the gastric and intestinal mucosa, by the cells of the islets of Langerrhans. There are five known somatostatin receptors which when activated by the ligand caused an inhibition of gastric acid secretion, pancreatic and biliary secretions. The somatostatin analogues have different vascular effects documented as downregulation of VEGF expression or decreasing the splanchnic flow.

Thus, the somatostatin analogs can have an effect on the prevention of rebleeding secondary to angiodysplasia by several mechanisms: inhibition of angiogenesis, reduction of splanchnic blood flow, increased vascular resistance and increased platelet aggregation.

Several cohort studies suggest that treatment with somatostatin analogues, octreotide can reduce the need for transfusion in patients with recurrent bleeding due to angiodysplasia. A meta-analysis of these studies, which included 62 patients in total found a relative risk of rebleeding of 0.76 (95% CI: 0.64 to 0.85) and a decrease of 2.2 transfusions (95% : -3.9 to -0.5) between the period before the treatment and the period of treatment with octreotide.

To date, there are no randomized phase III study to suggest the efficacy of somatostatin analogues in the prevention of rebleeding due to angiodysplasia.

Pasireotide is a new analogue of somatostatin which has a higher affinity of Octreotide to like receptors 1, 3 and 5. A preliminary study showed that pasireotide could be effective in the symptomatic treatment of endocrine tumors beyond the octreotide therapy. This superior efficacy of pasireotide compared to Octreotide justifies the evaluation pasireotide in the prevention of rebleeding due to angiodysplasia. Side effects described with the LP pasireotide are the possibility of post prandial hyperglycemia transient dose-dependent. Episodes of intestinal disorders have been reported (diarrhea, nausea, vomiting), but usually require no medicinal treatment and disappearing spontaneously during treatment.

All these data suggests for a randomized study against placebo to establish the efficacy of treatment with pasireotide LP in the prevention of rebleeding due to angiodysplasia. A randomized phase II feasibility study will be conducted to verify the the investigators hypotheis and followed if necessary by a phase III study.

Somatostatin analogs have vascular action that has been shown in other pathologies (gastrointestinal bleeding in patients with portal hypertension). Cohort studies suggest efficacy in reduction of transfusion requirements in patients with gastrointestinal angiodysplasia. In case of failure of endoscopic treatment there is no currently licensed treatment for the prevention of rebleeding in these patients.

The investigators objective is to evaluate the reduction in the number of red blood cells transfused to M6 in patients treated with pasireotide LP or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Angiodysplasia of the stomach, small intestine or colon confirmed by endoscopy.
2. 6 or more of packed red cells unit transfusion during the 6 months prior inclusion.
3. Failed endoscopic therapy or cons-indication for endoscopic treatment.
4. Patient affiliated to a social security insurance.
5. Age > 18 years.
6. Consent signed by the patient.

Exclusion Criteria:

1. Treatment with somatostatin analogue in the 6 months prior to inclusion
2. Symptomatic cholelithiasis
3. Rendu-Osler disease
4. Uncontrolled diabetes (HbA1c > 8%)
5. Breaking of the esophageal varicose veins bleeding older than six months.
6. Patients treated with anti vitamin K at baseline and during the study.
7. Patients with (AST, ALT> 2 ULN) and / or total bilirubin > 1.5 ULN.
8. TP < 50%, platelets <75 000/mm3, aPTT> 1.5 times the control
9. Uncontrolled heart disease: myocardial infarction within 6 months, status epilepticus angina, congestive heart failure grade III and NYHA, ventricular tachycardia, ventricular fibrillation, heart block, severe
10. Family medical history of the idiopathic sudden death
11. Syncope like medical history
12. QTcF> 450 ms
13. Metastatic malignancy
14. Pregnant or nursing women, women of childbearing age who have not achieved pregnancy test, women and men of reproductive age without effective contraception
15. Impossible follow for psychological and/or geographical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
number of red blood cells transfused | at 6 months
  number of red blood cells transfused at 6 months in patients treated with pasireotide or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, Principal Investigator — Société Française d'Endoscopie Digestive
Locations (1):
- Société Française d'Endoscopie Digestive (SFED), Paris, France

REFERENCES:
- [Background] Boley SJ, Sammartano R, Adams A, DiBiase A, Kleinhaus S, Sprayregen S. On the nature and etiology of vascular ectasias of the colon. Degenerative lesions of aging. Gastroenterology. 1977 Apr;72(4 Pt 1):650-60. PMID 300063
- [Background] Foutch PG, Rex DK, Lieberman DA. Prevalence and natural history of colonic angiodysplasia among healthy asymptomatic people. Am J Gastroenterol. 1995 Apr;90(4):564-7. PMID 7717311
- [Background] Vreeburg EM, Snel P, de Bruijne JW, Bartelsman JF, Rauws EA, Tytgat GN. Acute upper gastrointestinal bleeding in the Amsterdam area: incidence, diagnosis, and clinical outcome. Am J Gastroenterol. 1997 Feb;92(2):236-43. PMID 9040198
- [Background] Ohmiya N, Yano T, Yamamoto H, Arakawa D, Nakamura M, Honda W, Itoh A, Hirooka Y, Niwa Y, Maeda O, Ando T, Yao T, Matsui T, Iida M, Tanaka S, Chiba T, Sakamoto C, Sugano K, Goto H. Diagnosis and treatment of obscure GI bleeding at double balloon endoscopy. Gastrointest Endosc. 2007 Sep;66(3 Suppl):S72-7. doi: 10.1016/j.gie.2007.05.041. PMID 17709039
- [Background] Chalasani N, Cotsonis G, Wilcox CM. Upper gastrointestinal bleeding in patients with chronic renal failure: role of vascular ectasia. Am J Gastroenterol. 1996 Nov;91(11):2329-32. PMID 8931412
- [Background] Bhutani MS, Gupta SC, Markert RJ, Barde CJ, Donese R, Gopalswamy N. A prospective controlled evaluation of endoscopic detection of angiodysplasia and its association with aortic valve disease. Gastrointest Endosc. 1995 Nov;42(5):398-402. doi: 10.1016/s0016-5107(95)70038-2. PMID 8566626
- [Background] Veyradier A, Balian A, Wolf M, Giraud V, Montembault S, Obert B, Dagher I, Chaput JC, Meyer D, Naveau S. Abnormal von Willebrand factor in bleeding angiodysplasias of the digestive tract. Gastroenterology. 2001 Feb;120(2):346-53. doi: 10.1053/gast.2001.21204. PMID 11159874
- [Background] Pavey DA, Craig PI. Endoscopic therapy for upper-GI vascular ectasias. Gastrointest Endosc. 2004 Feb;59(2):233-8. doi: 10.1016/s0016-5107(03)02539-2. PMID 14745397
- [Background] Junquera F, Feu F, Papo M, Videla S, Armengol JR, Bordas JM, Saperas E, Pique JM, Malagelada JR. A multicenter, randomized, clinical trial of hormonal therapy in the prevention of rebleeding from gastrointestinal angiodysplasia. Gastroenterology. 2001 Nov;121(5):1073-9. doi: 10.1053/gast.2001.28650. PMID 11677198
- [Background] Bauditz J, Lochs H, Voderholzer W. Macroscopic appearance of intestinal angiodysplasias under antiangiogenic treatment with thalidomide. Endoscopy. 2006 Oct;38(10):1036-9. doi: 10.1055/s-2006-944829. PMID 17058171
- [Background] Dabak V, Kuriakose P, Kamboj G, Shurafa M. A pilot study of thalidomide in recurrent GI bleeding due to angiodysplasias. Dig Dis Sci. 2008 Jun;53(6):1632-5. doi: 10.1007/s10620-007-0067-z. PMID 17990111
- [Background] Kurosaki M, Saegert W, Abe T, Ludecke DK. Expression of vascular endothelial growth factor in growth hormone-secreting pituitary adenomas: special reference to the octreotide treatment. Neurol Res. 2008 Jun;30(5):518-22. doi: 10.1179/174313208X289499. PMID 18953743
- [Background] Ludwig D, Terai S, Bruning A, Stange EF. Long-term haemodynamic effects of octreotide on postprandial splanchnic hyperemia in humans: a placebo-controlled echo-doppler study. Aliment Pharmacol Ther. 1999 Aug;13(8):1119-29. doi: 10.1046/j.1365-2036.1999.00583.x. PMID 10468691
- [Background] Szilagyi A, Ghali MP. Pharmacological therapy of vascular malformations of the gastrointestinal tract. Can J Gastroenterol. 2006 Mar;20(3):171-8. doi: 10.1155/2006/859435. PMID 16550261
- [Background] Nardone G, Rocco A, Balzano T, Budillon G. The efficacy of octreotide therapy in chronic bleeding due to vascular abnormalities of the gastrointestinal tract. Aliment Pharmacol Ther. 1999 Nov;13(11):1429-36. doi: 10.1046/j.1365-2036.1999.00647.x. PMID 10571598
- [Background] Scaglione G, Pietrini L, Russo F, Franco MR, Sorrentini I. Long-acting octreotide as rescue therapy in chronic bleeding from gastrointestinal angiodysplasia. Aliment Pharmacol Ther. 2007 Sep 15;26(6):935-42. doi: 10.1111/j.1365-2036.2007.03435.x. PMID 17767478
- [Background] Brown C, Subramanian V, Wilcox CM, Peter S. Somatostatin analogues in the treatment of recurrent bleeding from gastrointestinal vascular malformations: an overview and systematic review of prospective observational studies. Dig Dis Sci. 2010 Aug;55(8):2129-34. doi: 10.1007/s10620-010-1193-6. PMID 20393879
- [Background] Weckbecker G, Briner U, Lewis I, Bruns C. SOM230: a new somatostatin peptidomimetic with potent inhibitory effects on the growth hormone/insulin-like growth factor-I axis in rats, primates, and dogs. Endocrinology. 2002 Oct;143(10):4123-30. doi: 10.1210/en.2002-220219. PMID 12239124